CLINICAL TRIAL: NCT05979480
Title: The Effects of Growth Hormone Treatment Discontinuation in Adults on Metabolic Profile, Body Composition and Quality Of Life
Brief Title: The Effects of Growth Hormone Treatment Discontinuation in Adults on Metabolic Profile, Body Composition and Quality Of Life (GAMBOL Study)
Acronym: GAMBOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: RRK7819
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Growth Hormone Treatment Continuation Group: Adult patients with GHD who have been on GH treatment for at least 5 years and will be continuing their treatment whilst on the study.
  Interventions: Diagnostic Test: Dual energy X-ray absorptiometry (DXA)
- Growth Hormone Treatment Discontinuation Group: Adult patients with GHD who have been on GH treatment for at least 5 years and will be discontinuing their treatment whilst on the study for 2 years.
  Interventions: Diagnostic Test: Dual energy X-ray absorptiometry (DXA)

INTERVENTIONS:
Diagnostic Test: Dual energy X-ray absorptiometry (DXA) — DXA scan to assess bone mineral density, fat mass and muscle mass.

SUMMARY:
Background Growth hormone (GH) is a hormone produced by the pituitary gland which sits at the base of the brain. In adults, GH plays an important role in keeping the bones and muscles healthy, and in regulating the levels of sugar and fat in the body. Growth hormone deficiency (GHD) is a condition where the pituitary gland does not make as much GH as the body needs. The most common cause is damage to the pituitary gland due to tumours (growth), surgery or radiotherapy. In the UK, around 1 in 10,000 adult people have GHD. If left untreated, adults with GHD may experience tiredness and low mood, develop weaker bones, have increased body fat and high cholesterol.

Research has shown that treatment with daily GH injections can improve the symptoms experienced by patients with GHD, but the beneficial effects of GH treatment have only been studied over a short period of 4 to 12 months. In the UK, most adults with GHD are prescribed with GH indefinitely. Some adult patients, who have been on GH treatment for a long time, have wondered what would happen if they stopped taking GH. Will their symptoms come back or not? At the moment, there is no research evidence that clearly answer this question. Hence, a systematic investigation is urgently needed to examine what happens when adult patients with GHD stop taking GH.

Aims The main aim of this study is to establish if it would be feasible to conduct a robust and systematic study called a randomised control trial (RCT), to compare the effects of continuing and stopping long-term GH treatment in adult patients with GHD. This study will: (1) assess whether patients taking GH injection, would agree to take part in a study involving stopping their GH injection and being monitored over a period of time and (2) whether patients would be willing to stop or continue their GH injections by chance (random selection) if accepted in the study.

Methods

This project includes three separate studies:

* Phase 1: Online national survey of UK GHD specialists treating adult patients with GHD.
* Phase 2: Feasibility study involving two groups of adult patients with GHD who have been receiving GH treatment for at least 5 years. Patients will be recruited from two GHD specialist centres in Birmingham. One group (intervention) will include 20-25 patients who are willing to stop taking GH treatment for 2 years. The second group (control) will include 20-25 patients who wish to continue their GH treatment and are willing to undergo monitoring for 2 years. The monitoring will involve blood tests and completing quality of life questionnaires every 6 months, and measurements of body fat, muscles mass and bone mineral density at the beginning and at the end of the study.
* Phase 3: Face-to-face or telephone interviews with 10-16 patients to explore in detail their experiences of participating, completing and/or withdrawing from the study.

Patient and Public Involvement A patient and public advisory group has helped design this proposal and will be involved throughout the research project. The group will review the study protocol, help develop the necessary information resources for participants and assist with interpretation of the results.

Dissemination The results of the study will be submitted for publication in medical journals in the field of GHD. The results will also be presented at the Pituitary Foundation meetings and at local, national and international conferences. Members of the patient and public advisory group will also help in sharing the information about the study with the wider public through relevant charities and social media.

DETAILED DESCRIPTION:
1. BACKGROUND

   Growth hormone deficiency (GHD) in adults is caused by decreased secretion of growth hormone (GH) from the pituitary gland (1, 2). This condition is usually caused by a tumour, surgery and/or radiotherapy involving the pituitary gland (3). Adults with GHD present with a constellation of several non-specific features including low mood, poor general well-being, reduced bone mineral density (BMD), increased body fat, increased cholesterol level and reduced exercise capacity (3, 4, 5). Treatment with recombinant human growth hormone (GH) injection has been proven, in short-term studies, to improve the wide spectrum of health issues associated with GHD (6).

   In the UK, the National Institute for Health and Care Excellence (NICE) recommends treating adult patients with GHD with GH until peak bone and muscle mass have been achieved (estimated to be at around the age of 25 years) (7) . For adults over 25 years old, the prescribing of GH treatment is based on the NICE criteria which requires patients to: a) have severe GHD, defined as peak GH response of less than 9 mU/litre during a GH stimulation test; b) have a perceived impairment of quality of life (QoL), as demonstrated by a score of at least 11 in the 'Quality of Life - Adult Growth Hormone Deficiency Assessment' (QoL-AGHDA) questionnaire; c) be receiving appropriate treatment for any other pituitary hormone deficiencies. The UK population of adult patients with GHD receiving GH is quite unique and homogenous as they all have severe GHD and poor quality of life (QoL) prior to commencing the treatment (4). The UK is the only country in the world that offers GH to adult patients with GHD only after poor QoL scores have been confirmed by using the QoL-AGHDA questionnaire (1, 4, 6).

   In the UK, provided that a 7-point improvement (or higher) on the 25-point QoL-AGHDA scale is demonstrated during the first 9 months of GH therapy, adult patients with GHD can continue with their GH treatment long-term (7). However, it remains uncertain if the beneficial effects of GH therapy are sustained throughout adult life, as robust evidence on the risks and benefits of long-term GH treatment is limited. Furthermore, the evidence of improved QoL in adult patients with GHD having GH treatment over placebo has not been established (6). Anecdotally, clinicians report encountering patients who question the merit of continuing with long-term GH treatment. Paradoxically, the same patients are apparently reluctant to stop GH therapy due to fears of return of symptoms and uncertainty about the short-term and long-term effects of treatment discontinuation. Consequently, and in the absence of clear evidence and definitive guidance, replacement therapy with GH continues indefinitely in many adults.

   To date, the optimal duration of GH replacement therapy in adults and the consequences of treatment withdrawal have not been established. There are only few, mainly short-term, follow-up studies which, however, provide conflicting results. Overall, the beneficial effects of GH treatment appear to occur during the first year of therapy with only a few studies reporting sustained benefits up to 5 years (5, 8-10). It is well established that GH secretion decreases with advancing age and that low GH levels are even associated with increased longevity and decreased morbidity (11, 12). Currently, many adults with GHD are receiving GH indefinitely without knowing if continuing or discontinuing long-term treatment has sustained beneficial or even adverse effects (13, 14). Similarly, reliable data on the impact of discontinuing long-term GH therapy in adults is practically not available.
2. RATIONALE

   Many questions on the effectiveness of long-term treatment with GH in adults remain unanswered including its optimal duration and the consequences of treatment discontinuation. The primary aim of this study is to assess the feasibility of conducting a large-scale multi-centre study to evaluate the effects of discontinuation of long-term GH therapy on the metabolic profile, body composition and QoL in a cohort of adult patients with GHD (aged 25 years and over) over a period of 24 months.

   Currently, much of the evidence on safety-related issues associated with long-term GH therapy comes from uncontrolled retrospective, and observational studies, which are methodologically inferior compared with randomised control trial (RCT) (1, 6). A critical assessment of data from limited RCTs did not show consistent beneficial effects of GH therapy in adult patients with GHD compared with placebo (6). In 2016, several international endocrine societies collectively highlighted the need for carefully designed and rigorously conducted cohort studies to monitor the safety of long-term GH therapy (15). Furthermore, treatment of adults with GHD is also associated with significant health care costs. In the UK, the average annual cost of GH treatment in adults is estimated to be around £3,350 per patient, with a life-long therapy cost of between £42,000 and £45,400 (7). Furthermore, the treatment regimen of daily self-injections can be inconvenient and burdensome for many patients (14, 16).

   The current NICE guidance provides clear criteria for commencing GH treatment for adults with GHD. However, it but does not offer any recommendations on the optimal duration of GH treatment in adults or if and when discontinuation should be considered. Consequently, GH replacement therapy tends to be offered indefinitely even when patients fail to report any sustained benefits from this treatment. Given that GH treatment is associated with significant health care costs, it is imperative to clearly establish the clinical and cost-effectiveness of the therapy. A methodologically robust and well-designed large-scale multi-centre study will contribute this evidence. However, Medical Research Council guidelines suggest that feasibility studies are required to test the methodology and establish the specific parameters prior to any full large-scale multi-centre study (17). The strict criteria for prescribing GH to adults and the homogeneity of the UK population of adults with GHD, offers an ideal setting to undertake a robust study.
3. THEORETICAL FRAMEWORK

   In clinical practice, some patients question the merit of continuing their long-term GH treatment due to the subjective perceived lack of benefits. Currently, there are no guidelines informing the optimal duration of GH therapy in adults. As a result, GH is prescribed indefinitely without clear evidence on the benefits of long-term treatment. Undoubtedly, an RCT comparing continuation versus discontinuation of long-term GH therapy is needed to understand the impacts of treatment discontinuation in adults. However, prior to embarking on an RCT, the feasibility of a discontinuation study and the acceptability of randomisation to patients and clinicians need to be assessed.

   In 2018, NHS England stated that 'new research should only be undertaken in areas where there is a defined evidence gap and the need for the research can be clearly articulated, and this project accords with that principle (18). The strict criteria for prescribing GH to adults and the homogeneity of the UK population of adults with GHD, offers an ideal setting to undertake a robust study. A methodologically robust and well-designed large-scale multi-centre study will contribute this evidence. However, Medical Research Council guidelines suggest that feasibility studies are required to test the methodology and establish the specific parameters prior to any full large-scale multi-centre study (17).
4. RESEARCH QUESTION/AIM(S)

   The primary aim of this study is to assess the feasibility of conducting a large-scale multi-centre study that will evaluate the effects of discontinuation of long-term GH therapy on the metabolic profile, body composition and QoL in a cohort of adult patients with GHD (aged 25 years and over) over a period of 24 months. In the conduct of this study, the following questions are anticipated to be answered:
   * Is it feasible to conduct a large multi-centre study on the effects of discontinuation of long-term GH treatment in adults?
   * Is it feasible to recruit and retain patients into the study?
   * What are the factors influencing recruitment, retention and drop out?
   * What are the patients' views about being randomised into a discontinuation or a continuation group?

   4.1 Objectives

   The main objectives of this study are:
   1. Phase 1: to understand the current practice of endocrine clinicians in the UK of offering GH treatment discontinuation in adults with GHD who have been on long-term replacement therapy. It will also determine the willingness of endocrine clinicians in the UK to take part in a future large-scale multi-centre study;
   2. Phase 2: to assess the feasibility of conducting a large-scale multi-centre study on discontinuation of long-term GH treatment in adult patients with GHD;
   3. Phase 3: to explore the experiences of participants in completing and/or withdrawing from the study, to identify barriers to recruitment and retention and explore participants' views about the use of randomisation in future large-scale multi-centre study.

   4.2 Outcome

   Answering the primary objectives of this study will help assess the feasibility of future large-scale multi-centre study. The primary outcome measures from the phase 2 and phase 3 of the study will include:
   1. Consent rate
   2. Completion rate
   3. Withdrawal rate
   4. Adverse events

   Additionally, the following secondary outcome measures are expected from the study:
   1. Measurement of anthropometric parameters (height, weight, body mass index [BMI], blood pressure, waist and hip circumferences), lipids profile, glycated haemoglobin A1c (HbA1c) and body composition (bone mineral density [lumbar spine and both hips], fat mass and muscle mass using dual-energy X-ray absorptiometry [DXA] scan) over a period 24 months;
   2. Barriers for recruiting and retaining participants into the study;
   3. Suitability and acceptability for patients of the frequency of follow-up and assessment;
   4. Suitability and acceptability for patients of the QoL questionnaires;
   5. Suitability of the study protocol including recruitment, biochemical monitoring, body composition monitoring and QoL assessment;
   6. Safety of growth hormone treatment discontinuation in adult patients with GHD.
5. STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYIS

This is a sequential mixed-methods study which will be conducted in three phases:

* (Phase 1) Survey of endocrine clinicians (Ethics approval is not being sought for this part of the study as it is not required. Details provided are for information only)
* Phase 2: Observational feasibility cohort study
* Phase 3: Qualitative study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25 years and over with GHD.
* GHD previously confirmed by a validated test as per guideline (7).
* On GH replacement therapy for 5 years or longer.
* Able to provide informed written consent.

Exclusion Criteria:

* Patients with poorly controlled diabetes (defined as having an HbA1c of >7%), poorly controlled hyperlipidaemia and severe cardiovascular disease.
* Patients receiving treatment for low BMD or deemed to be requiring treatment for low BMD during baseline screening.
* Patients who are unable to provide informed written consent.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve two groups of adult patients with GHD (aged 25 years and over).
  * Discontinuation group: 20-25 patients who have been on GH therapy for 5 years or longer and voluntarily agree to discontinue their treatment and be monitored for 2 years.
  * Continuation group: 20-25 patients who have been on GH therapy for 5 years or longer and voluntarily agree to take part in the study where their treatment is continued and are monitored in the same way as the discontinuation group.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Consent Rate | June 2025
Complete Rate | August 2025
Withdrawal Rate | August 2025
Adverse Events | August 2025

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share patient data to other researchers